CLINICAL TRIAL: NCT02247063
Title: Motor Cortex as a Research and Therapeutic Target in TMD
Brief Title: Motor Cortex as a Research & Therapeutic Target in TMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Alexandre DaSilva, DDS, DMedSc, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 70766
Record Dates: First submitted 2014-09-18; First posted 2014-09-23 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Sham Comparator): The subjects in the placebo arm will participate in 5 daily M1 High-Definition Transcranial Direct Current Stimulation (HD-tDCS) sessions. During each session, a modular EEG recording cap will be placed on the subject's head and the anodal electrode will be placed on the motor cortex contralateral to the worst TMD pain side (C3). Current will be applied only for 30 seconds - this is a reliable method of sham stimulation (Gandiga et al., 2006) as sensations arising from tDCS treatment occur only at the beginning of application.
  Interventions: Device: High-Definition Transcranial Direct Current Stimulation (HD-tDCS)
- Experimental (Experimental): The subjects in the experimental arm will participate in 5 daily sessions. During each session, a modular EEG recording cap will be placed on the subject's head and the anodal electrode will be placed on the motor cortex contralateral to the worst TMD pain side (C3). Then 2mA of transcranial direct current stimulation will be applied for 20 minutes.
  Interventions: Device: High-Definition Transcranial Direct Current Stimulation (HD-tDCS)

INTERVENTIONS:
Device: High-Definition Transcranial Direct Current Stimulation (HD-tDCS) — HD-tDCS is a non-invasive brain neuromodulatory method for M1 that involves sending a weak electrical current into your brain.

SUMMARY:
The investigators are doing a study to learn about the effects of a type of low-energy non-surgical electrical brain stimulation (HD-tDCS) on chronic pain in people's jaw joints. Disorders in these joints are called temporomandibular joint disorders, or TMD.

DETAILED DESCRIPTION:
Chronic temporomandibular joint disorders (TMD) represent clinical problems in which empirical treatments offer uncertain relief for a large number of patients. Many conventional therapies are ineffectual, leading to persistent treatment failure and/or poor iatrogenic-induced results; which raises the possibility that the cause for their pain endurance may also lie in the brain milieu. Although MRI-based techniques have provided insights into some neuroplastic mechanisms of TMD in humans, many questions regarding its molecular mechanisms in vivo are still unanswered. First, how are endogenous μ-opioid mechanisms in the brain, known to be centrally involved in pain regulation, affected by acute and chronic TMD pain? Second, how can they be directly modulated to provide analgesic effect on pain measures? Finally, what are the neuroplastic effects in the brain after continuous modulation of those molecular mechanisms? The understanding of these processes is crucial to determine the mechanisms engaged in the persistence and, most important, the alleviation of TMD.

Preliminary studies from our center, using positron emission tomography (PET) with [11C] carfentanil, a selective radiotracer for mu-opioid receptor (muOR), have demonstrated that there is a decrease in μOR availability (non-displaceable binding potential -BPND) in key pain-related structures in the brains of chronic trigeminal pain patients, which correlated with their clinical pain measures. We propose to demonstrate that acute (masseteric pain challenge) and chronic clinical pain measures in TMD patients are correlated with μ-opioid receptor (µOR) non-displaceable binding potential (BPND) in the thalamus and other pain-related regions.

ELIGIBILITY:
Inclusion Criteria:

* Daily chronic TMD pain and dysfunction for at least one year (Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) Axis I Group I: Myofascial pain diagnosis[15]) not adequately controlled by previous conventional therapies (TMJ open-surgery naïve) for more than

  1 year
* Self-reported pain score of at least 3 on a 0-10 scale in spite of existing treatment in the two weeks preceding the onset of the study
* Taking stable doses of medications for at least 4 weeks (if taking medications), and willing to limit the introduction of new medications for chronic TMD symptoms during the study

Exclusion Criteria:

* Pain not primarily due to TMD
* History or current evidence of a psychotic disorder (e.g. schizophrenia) or substance abuse by DSM-IV criteria; bipolar or severe major depression
* History of neurological disorder (e.g. epilepsy, stroke, neuropathy, neuropathic pain)
* Any severe clinical condition that in the opinion of the principal investigator interferes with the study
* Pregnant or expecting to become pregnant during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre FM DaSilva, DDS, DMedSc, Principal Investigator — University of Michigan

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: The subjects in the placebo arm will participate in 5 daily M1 High-Definition Transcranial Direct Current Stimulation (HD-tDCS) sessions. During each session, a modular EEG recording cap will be placed on the subject's head and the anodal electrode will be placed on the motor cortex contralateral to the worst TMD pain side (C3). Current will be applied only for 30 seconds - this is a reliable method of sham stimulation (Gandiga et al., 2006) as sensations arising from tDCS treatment occur only at the beginning of application.
  High-Definition Transcranial Direct Current Stimulation (HD-tDCS): HD-tDCS is a non-invasive brain neuromodulatory method for M1that involves sending a weak electrical current into your brain.
- Experimental: The subjects in the experimental arm will participate in 5 daily sessions. During each session, a modular EEG recording cap will be placed on the subject's head and the anodal electrode will be placed on the motor cortex contralateral to the worst TMD pain side (C3). Then 2mA of transcranial direct current stimulation will be applied for 20 minutes.
  High-Definition Transcranial Direct Current Stimulation (HD-tDCS): HD-tDCS is a non-invasive brain neuromodulatory method for M1that involves sending a weak electrical current into your brain.
Period: Overall Study
Arm/Group | Placebo | Experimental
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Experimental | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (16.7) | 34.8 (13.7) | 35.2 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pain Relief as Measured by Visual Analog Scale (VAS) Decrease of 50% or Greater From Baseline
Description: Self-reported VAS from 0 (no pain) to 10 (worst possible pain)
Time Frame: Post tDCS sessions compared to baseline (one week)
Measure: Number; unit: participants
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 12 | 12
participants | 4 | 9

2. Secondary Outcome: Number of Participants With Pain Relief as Measured by Visual Analog Scale (VAS) Decrease of 50% or Greater From Baseline
Description: Self-reported VAS from 0 (no pain) to 10 (worst possible pain)
Time Frame: One month after tDCS sessions compared to baseline (6 weeks)
Measure: Number; unit: participants
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 12 | 12
participants | 4 | 9

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Placebo | Experimental
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Experimental (N=12)
Headache (General disorders) | 8 | 7
Neck Pain (General disorders) | 8 | 8
Scalp Pain (General disorders) | 10 | 8
Scalp Burn (Sensation) (General disorders) | 4 | 6
Tingling (General disorders) | 11 | 10
Skin Redness (General disorders) | 1 | 2
Sleepiness (General disorders) | 10 | 9
Trouble Concentrating (General disorders) | 9 | 3
Mood Change (General disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes